CLINICAL TRIAL: NCT02879942
Title: First-trimester Study of the Morphometric Characteristics of the Placenta to Assess the Risk of Preeclampsia and Intrauterine Growth Restriction in Singleton Pregnancies
Brief Title: First Trimester Placental Assessment in the Screening of Preeclampsia and Intrauterine Growth Restriction
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Other Study IDs: IIBSP-PLA-2016-31
Record Dates: First submitted 2016-07-20; First posted 2016-08-26 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Preeclampsia; Intrauterine Growth Restriction
Keywords: Placental volume; First-trimester screening; Ultrasound; Preeclampsia; Intrauterine growth restriction; Biochemical markers; Uterine artery doppler
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples from the first blood test performed during pregnancy

GROUPS / COHORTS (2):
- Case cohort: Patients with pregnancies complicated by placental insufficiency (preeclampsia and/or intrauterine growth restriction) will be included in this cohort.
  Interventions: Other: Ultrasound study of the placenta; Other: Measurement of angiogenic and anti-angiogenic factors (sFlt-1 and PlGF) in the first trimestre blood test
- Control cohort: Patients with pregnancies not complicated by placental insufficiency (preeclampsia and/or intrauterine growth restriction) will be included in this cohort.
  Interventions: Other: Ultrasound study of the placenta; Other: Measurement of angiogenic and anti-angiogenic factors (sFlt-1 and PlGF) in the first trimestre blood test

INTERVENTIONS:
Other: Ultrasound study of the placenta — The placenta will be scanned to measure the placental volume, chorionic plate, basal plate and thickness.
Other: Measurement of angiogenic and anti-angiogenic factors (sFlt-1 and PlGF) in the first trimestre blood test

SUMMARY:
Preeclampsia (PE) and intrauterine growth restriction (IUGR) are clinical manifestations of placental insufficiency. These complications affect 5-15% of pregnancies, and are responsible for up to 20% of preterm births. Women who develop PE during pregnancy also have an increased risk for cardiovascular events, both at short and long term. This justifies the need to improve diagnostic tools to identify patients at risk for these complications. PE and IUGR are multifactorial entities. Screening algorithms should thus include several parameters to achieve high detection rates. Research has mainly focused in the analysis of biophysical and biochemical parameters, and the study of the placenta itself has not been included in current diagnostic strategies. Investigators hypothesize that detection rates of preeclampsia and intrauterine growth restriction could be improved by the study of placental characteristics in the first trimester of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* pregnancies with fetuses with CRL between 45 and 80mm
* absence of chromosomal abnormalities
* absence of congenital anomalies
* absence of congenital infections

Exclusion Criteria:

* patient not accepting to participate in the study
* multiple pregnancies
* pregnancies without ultrasonographic confirmation of gestational age

Ages: 11 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with singleton pregnancies and ultrasonographic evaluation between 11+0 and 13+6 weeks of gestation
Sampling Method: Non-Probability Sample
Enrollment: 1390 (Actual)
Dates: Start 2016-08; Primary Completion 2020-02 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Development of preeclampsia | Up to birth
  Pre-eclampsia is diagnosed after 20 week of gestation with systolic blood pressure equal to or greater than 140 mmHg, diastolic blood pressure equal to or greater than 90 mmHg and proteinuria greater than or equal 0.3 g/d by 24 hour urine collection
Development of intrauterine growth restriction | At birth
  Intrauterine growth restriction is defined as birthweight below 10th centile according to local standards

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Trilla, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain